CLINICAL TRIAL: NCT05121506
Title: A Single-arm Open-label Study to Investigate the Bioavailability and Skin Absorption of CBD and THC From GT4 Technology in Healthy Adults
Brief Title: A Study to Investigate the Bioavailability and Skin Absorption of CBD and THC From GT4 Technology in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gefion Canada Inc. (Other)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19GBHG
Record Dates: First submitted 2021-11-04; First posted 2021-11-16 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Biological Availability; Skin Absorption; CBD; THC
Keywords: CBD; THC; GT4 Technology
MeSH Terms: interventions — Dronabinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBD and THC with GT4 technology (Experimental)
  Interventions: Combination Product: CBD and THC with GT4 technology

INTERVENTIONS:
Combination Product: CBD and THC with GT4 technology — A single topical dose of CBD and THC will be administered with GT4 technology. The material will be provided in a single use pre-filled syringe.

SUMMARY:
The bioavailability of cannabinoids differs greatly for different routes of administration. When applied topically to the skin, they are absorbed through the skin or hair follicles while interacting with receptors to provide localized effects. To gain more information on the potential of this route of administration in therapeutic applications, this open-label study will investigate the skin absorption and bioavailability of CBD and THC delivered trans-dermally.

DETAILED DESCRIPTION:
The global use of cannabis for both recreational and medical purposes has deep historical origins. Medicinal cannabis has traditionally been used to treat nausea, inflammation, vomiting and pain. The use of cannabis is widespread, with over 147 million people worldwide consuming cannabis annually ). While cannabis regulations for recreational use have traditionally followed the prohibitionist model, Canadian legalization is expected to loosen the barriers to access and research of its potential medicinal and therapeutic benefits.

Cannabidiol (CBD) and Δ9-tetrahydrocannabinol (THC) are two naturally occurring phytocannabinoids found in cannabis. THC is the main psychoactive compound of cannabis and gives users a distinguished "high" feeling, whereas CBD studies have shown it does not have any mind-altering effects. Differences in molecular interactions and structural properties are responsible for the varied pharmacological effects of THC and CBD. Both Δ9-THC and CBD exert their effects by interacting with the receptors of the endocannabinoid system (ECS), CB1 and CB2, with varying affinities.

The ECS plays an integral role in regulatory functions implicated in health and disease as well as in downregulating stress signals that cause pain and inflammation. Endocannabinoid receptors are ubiquitous in the body, and due to their extensive presence, the ECS is referred to as a 'bridge between mind and body. Cutaneously, the role of the ECS is to regulate skin cell proliferation, survival, and differentiation. CB1 receptors are found mainly in the brain and central nervous system and are involved in coordination, movement, pain, memory and mood, whereas CB2 receptors are found mainly in peripheral organs and are linked with reducing inflammation, pain and tissue damage. Differential activation of CB1 and CB2 receptors, whether individually or simultaneously, could lead to varied physiological effects.

The differences in neurological outcomes between THC and CBD may be linked to their contrasting interactions with the CB1 receptor. THC is a potential partial agonist of the CB1 receptor, and it produces its effects through direct binding. CBD, on the other hand, is a negative allosteric modulator of CB1 and it induces a conformational change to inhibit other agonists from binding. The binding of CB1 receptors is also responsible for the antinociceptive activity of THC, which makes it an effective analgesic agent. In addition, THC has been shown to improve food intake and weight gain in wasting conditions such as cancer, Crohn's disease and AIDS, as well as in the treatment of glaucoma, nausea, multiple sclerosis, epilepsy and inflammation in a series of preclinical and clinical studies. CBD, on the other hand, shows immense therapeutic potential without the psychoactive effects of THC. It has shown promise in the treatment of anxiety, epilepsy, schizophrenia, Parkinson's disease, Alzheimer's disease, multiple sclerosis and sleep management. Studies have shown that CBD and THC acting together can be more potent than their individual effects. Oral supplementation of THC alone is not as effective as their combination, which has been shown to significantly relieve neuropathic pain. CBD can also lower the psychoactive effects of THC and thus produce their combined benefits by enhancing THC tolerability.

The bioavailability of cannabinoids differs immensely for different routes of administration. When taken orally, CBD and THC are digested in the stomach and intestines. Further the CBD and THC will undergo first-pass metabolism after digestion. When taken sublingually, they bypass first-pass metabolism, which increases their bioavailabilities. When inhaled, CBD and THC are immediately absorbed through the lungs resulting in a faster response and higher bioavailability in comparison with oral products. When applied topically to the skin, they are absorbed through the epidermis or hair follicles while interacting with receptors to provide localized effects. A common route of administration for recreational purposes is inhalation through smoking as it yields very high concentrations rapidly, but this is not ideal due to risks such as toxicity and loss of activity through combustion. To take advantage of the lungs' efficient drug delivery and avoid the harm associated with smoking, inhalation can be achieved via aerosolization or vaporization. Systemically, the bioavailability of inhaled CBD using these two methods has been reported to be 31%, and the peak plasma concentration was reached within 10 minutes. The terminal half-life of CBD following inhalation was found to be 27-35 hours, following intravenous injection it was 18-33 hours and following oral administration it was 2-5 days. The terminal half-life of THC after inhalation was found to be 21-31 hours and following intravenous injection it was 24 hours. Bioavailability of oral CBD was found to be around 6%, and bioavailability for oral THC was shown to be 4-12%.

The pharmacokinetics of CBD and THC after transdermal administration have not been extensively studied. When applied with the GT4 technology, the CBD and THC are expected to be absorbed through the stratum corneum and other epidermal layers, the basement membrane and into the dermis rapidly. Once in the dermis CBD and THC can enter the capillary bed aided by increased blood flow and then the systemic circulation. In addition to avoiding the negative effects of inhalation, transdermal administration is superior to oral ingestion as this route provides a way to avoid gastrointestinal involvement and first pass metabolism. Further, transdermal delivery may generate more constant plasma levels. It can also be designed for targeted delivery where the IP and specific tissues within the cutaneous ECS can interact. Pharmaceuticals with the GT4 technology have had over 1,000 prescriptions filled in the United States to deliver 10% gabapentin and 5% naproxen sodium for treatment of severe muscular skeletal pain. This technology has allowed physicians to treat severe pain without or with significantly less opioids. To date, no adverse events have been reported.

The objective of this open-label study is to investigate the bioavailability and skin absorption of CBD and THC delivered using GT4 technology in a healthy adult population. Participants will be healthy men and women between the ages of 25-65 and will be occasional cannabis users. They will have used cannabis at least once in the past 6 months and 4 times in their lifetime but no more than 3 times per week. Participants must have experienced psychotropic effects related to cannabis without having severe adverse events. In the area of application, participants must not have received laser hair removal, shaved, or waxed within 14 days or have any acute or chronic skin diseases or dermatological conditions to avoid interfering with the test product. Participants must not be using medicinal cannabis. They must not be receiving any treatments that may confound results, such as prescribed medications, over-the-counter medications, supplements, and food/drinks that will interact with the test product or that contain CBD and THC. Based on the short half lives of CBD and THC, recreational users must refrain from cannabis for 48 hours. The inclusion and exclusion criteria in this study ensure a homogeneous population of participants who are healthy, stable, and have no comorbidities.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females between 25-65 years of age at screening
2. Body Mass Index (BMI) from 18.5 to 29.9 kg/m2, inclusive
3. Occasional users of cannabis: Have consumed cannabis products at least once in the past 6 months and at least 4 times in their lifetime but no more than 3 times per week and not within 48 hours of Visit 2 and have experienced psychotropic effects without severe adverse events (short term paranoia, belligerence, extreme hallucinations) requiring medical interventions. Eligibility will be determined on a case by case basis by the QI
4. Female participant is not of child bearing potential, which is defined as females who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have undergone natural menopause (have not had menses for > 1 year) OR

   Females of childbearing potential must agree to abstain from heterosexual intercourse or use two methods of contraception for 30 days prior to first treatment and for 30 days after the treatment. Subjects must have a negative urine pregnancy test result at screening and baseline. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   1. Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   2. Double-barrier method
   3. Intrauterine devices
   4. Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   5. Vasectomy of partner at least 6- months prior to screening
5. A male participant with sexual partners who are not pregnant or do not fit the criteria as indicated above in number 4 must meet the following criteria

   * Participant is unlikely to procreate, defined as surgically sterile (i.e. has undergone vasectomy, it must be at least 6 months since the surgery)
   * Participant agrees to use of the accepted contraceptive regimens from first drug administration until 30 days after the drug administration
   * An acceptable method of contraception includes one of the following:

     * Abstinence from heterosexual intercourse
     * Condom with spermicide
6. Agrees to avoid alcohol intake 48 h prior to visit 2
7. Agrees to avoid tobacco or nicotine-containing products 96 hours prior to visit 2
8. Healthy as determined by medical history and laboratory results, as assessed by the QI
9. Agrees to complete all study related procedures and assessments
10. Agrees to provide information of two adult contacts to be reached in the event of transportation requirements from the clinic to their home after the study visits
11. Provides voluntary, written informed consent to participate in the study

Exclusion Criteria:

1. Women who are pregnant, breast feeding, or planning to become pregnant during the course of the trial
2. Allergy or sensitivity to investigational product's active or inactive ingredients
3. Acute or chronic skin disease (i.e. atopic dermatitis, eczema, rosacea, psoriasis) or dermatological conditions (open wounds, scars, sunburns, moles) in the proposed area of application that would interfere with the application and absorption of the test product
4. Shaving, waxing or laser hair removal of the planned study treatment application area within 14 days prior to baseline. Tattoos on the planned study application area.
5. Current use of prescribed medication containing the ingredients in the IP
6. Current use of over-the-counter medications, supplements, and foods/drinks containing the ingredients in the IP unless willing to washout
7. Prescribed or OTC medication, supplements, or food/drinks that will interact with the investigational product
8. Positive drug of abuse test at baseline
9. History of alcohol and/or drug abuse or substance dependence within the last 12 months
10. High alcohol intake (average of >2 standard drinks per day)
11. Self-reported serious psychological disorder(s) diagnosis e.g. schizophrenia, bipolar disorder, depression, PTSD, sleep disorder that, in the QI's opinion, could interfere with study participation. History of suicidal ideation, attempts and/or behaviour.
12. History of psychosis in immediate family including schizophrenia and affective psychosis
13. Cancer, except basal cell skin carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
14. Major surgery in the past 3 months or individuals who have planned surgery during the course of the trial. Participants with minor surgery will be considered on a case-by-case basis by the QI
15. Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
16. Self-reported cardiovascular disease. Participants with no significant cardiovascular event in the past 1 year and who are on stable medication may be included after assessment by the QI on a case-by-case basis
17. Individuals with an autoimmune disease or who are immune-compromised
18. Positive laboratory results for HIV, Hepatitis B or C as assessed at screening
19. Type I or Type II diabetes
20. Current or history of significant liver disease or dysfunction that in the opinion of the QI may impact study outcomes or participant safety
21. History of or current diagnosis with kidney diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones symptom-free for 6 months
22. Self-reported current or pre-existing thyroid condition. Treatment on a stable dose medication for over 6 months will be reviewed on a case-by-case basis by the QI
23. Self- reported blood/bleeding disorder as assessed by the QI
24. Clinically significant abnormal laboratory results at screening as determined by the QI
25. Blood donation 30 days prior to screening, during the study, or a planned donation within 30-days of the last study visit
26. Participation in other clinical research trials 30 days prior to enrollment will be assessed on a case-by-case basis by the QI
27. Individuals who are unable to give informed consent
28. Any other condition or lifestyle factor, that, in the opinion of the QI may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-11-27 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Area under the curve to the last measured timepoint (AUCT) for CBD metabolite following acute topical administration using GT4 technology of CBD and THC | 12-hour study period
  The AUCT will be calculated using the trapezoid approximation. Time points assessed for AUC0-12 h: pre-dose (T = 0 h) and post-dose at 10, 20, 30, 45 min and 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8 and 12 h.
Area under the curve to the last measured timepoint (AUCT) for THC metabolite following acute topical administration using GT4 technology of CBD and THC | 12-hour study period
  The AUCT will be calculated using the trapezoid approximation. Time points assessed for AUC0-12 h: pre-dose (T = 0 h) and post-dose at 10, 20, 30, 45 min and 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8 and 12 h. This parameter will be presented for each metabolite, for each study participant.
Maximum concentration (Cmax) for CBD metabolite following acute topical administration using GT4 technology of CBD and THC | 12-hour study period
  Peak concentration (Cmax) will be determined directly from the concentration-time curve.
Maximum concentration (Cmax) for THC metabolite following acute topical administration using GT4 technology of CBD and THC | 12-hour study period
  Peak concentration (Cmax) will be determined directly from the concentration-time curve.
Time to maximum concentration (Tmax) for CBD metabolite following acute topical administration using GT4 technology of CBD and THC | 12-hour study period
  Time to peak concentration (Tmax) will be determined directly from the concentration-time curve.
Time to maximum concentration (Tmax) for THC metabolite following acute topical administration using GT4 technology of CBD and THC | 12-hour study period
  Time to peak concentration (Tmax) will be determined directly from the concentration-time curve.
Area under the curve to infinity (AUCI) for CBD metabolite following acute topical administration using GT4 technology of CBD and THC | 12-hour study period
  The area under the curve to infinity AUCI will be calculated by AUCT + CT/ λ, where CT is the last quantifiable concentration.
Area under the curve to infinity (AUCI) for THC metabolite following acute topical administration using GT4 technology of CBD and THC | 12-hour study period
  The area under the curve to infinity AUCI will be calculated by AUCT + CT/ λ, where CT is the last quantifiable concentration.
Terminal elimination rate constant (λ or ke) for CBD metabolite following acute topical administration using GT4 technology of CBD and THC | 12-hour study period
  Terminal disposition rate constant (λ) will be calculated as the slope of points on the terminal log-linear end of the concentration versus time curve.
Terminal elimination rate constant (λ or ke) for THC metabolite following acute topical administration using GT4 technology of CBD and THC | 12-hour study period
  Terminal disposition rate constant (λ) will be calculated as the slope of points on the terminal log-linear end of the concentration versus time curve.
Terminal half-life (t1/2) for CBD metabolite following acute topical administration using GT4 technology of CBD and THC | 12-hour study period
  Terminal half-life (t1/2) will be calculated as ln(2)/λ = 0.693/λ.
Terminal half-life (t1/2) for THC metabolite following acute topical administration using GT4 technology of CBD and THC | 12-hour study period
  Terminal half-life (t1/2) will be calculated as ln(2)/λ = 0.693/λ.
Absorption rate constant (ka) for CBD metabolite following acute topical administration using GT4 technology of CBD and THC | 12-hour study period
  The absorption rate constant (ka) will be calculated using the feathering method.
Absorption rate constant (ka) for THC metabolite following acute topical administration using GT4 technology of CBD and THC | 12-hour study period
  The absorption rate constant (ka) will be calculated using the feathering method.

OTHER OUTCOMES:
Incidence of pre-emergent and post-emergent adverse events (AEs) following a single dose of CBD and THC from GT4 technology | 12-hour study period and follow-up call at 7 days
  Number of pre-emergent and post-emergent adverse events will be determined to calculate the incidence. Adverse events will be recorded during the 12 h in-clinic visit and during a follow-up phone call (7 days)
Change in Aspartate Aminotransferase at 12-h post dose following acute topical administration using GT4 technology of CBD and THC compared to baseline. | 12-hour study period
  Change in Aspartate Aminotransferase at 12-h post dose following acute topical administration using GT4 technology of CBD and THC will be compared to baseline.
Change in Alanine Aminotransferase at 12-h post dose following acute topical administration using GT4 technology of CBD and THC compared to baseline. | 12-hour study period
  Change in Alanine Aminotransferase at 12-h post dose following acute topical administration using GT4 technology of CBD and THC will be compared to baseline.
Change in Alkaline Phosphatase at 12-h post dose following acute topical administration using GT4 technology of CBD and THC compared to baseline | 12-hour study period
  Change in Alkaline Phosphatase at 12-h post dose following acute topical administration using GT4 technology of CBD and THC will be compared to baseline.
Change in Total Bilirubin at 12-h post dose following acute topical administration using GT4 technology of CBD and THC compared to baseline. | 12-hour study period
  Change in Total Bilirubin at 12-h post dose following acute topical administration using GT4 technology of CBD and THC will be compared to baseline.
Change in Creatinine at 12-h post dose following acute topical administration using GT4 technology of CBD and THC compared to baseline. | 12-hour study period
  Change in Creatinine at 12-h post dose following acute topical administration using GT4 technology of CBD and THC will be compared to baseline.
Change in Estimated Glomerular Filtration Rate (eGFR) at 12-h post dose following acute topical administration using GT4 technology of CBD and THC compared to baseline. | 12-hour study period
  Change in eGFR at 12-h post dose following acute topical administration using GT4 technology of CBD and THC will be compared to baseline.
Change in random glucose at 12-h post dose following acute topical administration using GT4 technology of CBD and THC compared to baseline. | 12-hour study period
  Change in random glucose at 12-h post dose following acute topical administration using GT4 technology of CBD and THC will be compared to baseline.
Change in sodium levels at 12-h post dose following acute topical administration using GT4 technology of CBD and THC compared to baseline. | 12-hour study period
  Change in sodium levels at 12-h post dose following acute topical administration using GT4 technology of CBD and THC will be compared to baseline.
Change in potassium levels at 12-h post dose following acute topical administration using GT4 technology of CBD and THC compared to baseline. | 12-hour study period
  Change in potassium levels at 12-h post dose following acute topical administration using GT4 technology of CBD and THC will be compared to baseline.
Change in chloride levels at 12-h post dose following acute topical administration using GT4 technology of CBD and THC compared to baseline. | 12-hour study period
  Change in chloride levels at 12-h post dose following acute topical administration using GT4 technology of CBD and THC will be compared to baseline.
Change in White Blood Cell Count (WBC) at 12-h post dose following acute topical administration using GT4 technology of CBD and THC compared to baseline. | 12-hour study period
  Change in WBC at 12-h post dose following acute topical administration using GT4 technology of CBD and THC will be compared to baseline.
Change in amount of Neutrophils at 12-h post dose following acute topical administration using GT4 technology of CBD and THC compared to baseline. | 12-hour study period
  Change in amount of Neutrophils at 12-h post dose following acute topical administration using GT4 technology of CBD and THC will be compared to baseline.
Change in amount of Lymphocytes at 12-h post dose following acute topical administration using GT4 technology of CBD and THC compared to baseline. | 12-hour study period
  Change in amount of Lymphocytes at 12-h post dose following acute topical administration using GT4 technology of CBD and THC will be compared to baseline.
Change in amount of Monocytes at 12-h post dose following acute topical administration using GT4 technology of CBD and THC compared to baseline. | 12-hour study period
  Change in amount of Monocytes at 12-h post dose following acute topical administration using GT4 technology of CBD and THC will be compared to baseline.
Change in amount of Eosinophils at 12-h post dose following acute topical administration using GT4 technology of CBD and THC compared to baseline. | 12-hour study period
  Change in amount of Eosinophils at 12-h post dose following acute topical administration using GT4 technology of CBD and THC will be compared to baseline.
Change in amount of Basophils at 12-h post dose following acute topical administration using GT4 technology of CBD and THC compared to baseline. | 12-hour study period
  Change in amount of Basophils at 12-h post dose following acute topical administration using GT4 technology of CBD and THC will be compared to baseline.
Change in Red Blood Cell Count (RBC) at 12-h post dose following acute topical administration using GT4 technology of CBD and THC compared to baseline. | 12-hour study period
  Change in Red Blood Cell Count (RBC) at 12-h post dose following acute topical administration using GT4 technology of CBD and THC will be compared to baseline.
Change in hemoglobin levels at 12-h post dose following acute topical administration using GT4 technology of CBD and THC compared to baseline. | 12-hour study period
  Change in hemoglobin levels at 12-h post dose following acute topical administration using GT4 technology of CBD and THC will be compared to baseline.
Change in hematocrit levels at 12-h post dose following acute topical administration using GT4 technology of CBD and THC compared to baseline. | 12-hour study period
  Change in hematocrit levels at 12-h post dose following acute topical administration using GT4 technology of CBD and THC will be compared to baseline.
Change in platelet count at 12-h post dose following acute topical administration using GT4 technology of CBD and THC compared to baseline. | 12-hour study period
  Change in platelet count at 12-h post dose following acute topical administration using GT4 technology of CBD and THC will be compared to baseline.
Change in Mean Corpuscular Volume (MCV) at 12-h post dose following acute topical administration using GT4 technology of CBD and THC compared to baseline. | 12-hour study period
  Change in MCV at 12-h post dose following acute topical administration using GT4 technology of CBD and THC will be compared to baseline.
Change in mean corpuscular hemoglobin (MCH) at 12-h post dose following acute topical administration using GT4 technology of CBD and THC compared to baseline. | 12-hour study period
  Change in MCH at 12-h post dose following acute topical administration using GT4 technology of CBD and THC will be compared to baseline.
Change in mean corpuscular hemoglobin concentration (MCHC) at 12-h post dose following acute topical administration using GT4 technology of CBD and THC compared to baseline. | 12-hour study period
  Change in MCHC at 12-h post dose following acute topical administration using GT4 technology of CBD and THC will be compared to baseline.
Change in red cell distribution width (RDW) at 12-h post dose following acute topical administration using GT4 technology of CBD and THC compared to baseline. | 12-hour study period
  Change in RDW at 12-h post dose following acute topical administration using GT4 technology of CBD and THC will be compared to baseline.
Psychoactive Assessment following acute topical administration using GT4 technology of CBD and THC. | 12-hour study period
  Psychoactive Assessment as administered at post-dose at 10, 20, 30, 45 min and 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8 and 12 h.
  The "Psychoactive Assessment" will be administered just before each post-dose blood draw with the following questions:
  1. Are you experiencing a "high" feeling?
  2. On a scale of 1 (least) to 10 (most), how intense is that feeling?
  3. Is this "high" feeling (other than intensity) different than past high experiences? If yes, please describe.
Area under the curve to the last measured timepoint (AUCT) for Cannabinol (CBN) metabolite following acute topical administration using GT4 technology of CBD and THC | 12-hour study period
  The AUCT will be calculated using the trapezoid approximation. Time points assessed for AUC0-12 h: pre-dose (T = 0 h) and post-dose at 10, 20, 30, 45 min and 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8 and 12 h.
Maximum concentration (Cmax) for Cannabinol (CBN) metabolite following acute topical administration using GT4 technology of CBD and THC | 12-hour study period
  Peak concentration (Cmax) will be determined directly from the concentration-time curve.
Time to maximum concentration (Tmax) for Cannabinol (CBN) metabolite following acute topical administration using GT4 technology of CBD and THC | 12-hour study period
  Time to peak concentration (Tmax) will be determined directly from the concentration-time curve.
Area under the curve to infinity (AUCI) for Cannabinol (CBN) metabolite following acute topical administration using GT4 technology of CBD and THC | 12-hour study period
  The area under the curve to infinity AUCI will be calculated by AUCT + CT/ λ, where CT is the last quantifiable concentration.
Terminal elimination rate constant (λ or ke) for Cannabinol (CBN) metabolite following acute topical administration using GT4 technology of CBD and THC | 12-hour study period
  Terminal disposition rate constant (λ) will be calculated as the slope of points on the terminal log-linear end of the concentration versus time curve.
Terminal half-life (t1/2) for Cannabinol (CBN) metabolite following acute topical administration using GT4 technology of CBD and THC | 12-hour study period
  Terminal half-life (t1/2) will be calculated as ln(2)/λ = 0.693/λ.
Absorption rate constant (ka) for for Cannabinol (CBN) metabolite following acute topical administration using GT4 technology of CBD and THC | 12-hour study period
  The absorption rate constant (ka) will be calculated using the feathering method.

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada

REFERENCES:
- [Derived] Varadi G, Zhu Z, Crowley HD, Moulin M, Dey R, Lewis ED, Evans M. Examining the Systemic Bioavailability of Cannabidiol and Tetrahydrocannabinol from a Novel Transdermal Delivery System in Healthy Adults: A Single-Arm, Open-Label, Exploratory Study. Adv Ther. 2023 Jan;40(1):282-293. doi: 10.1007/s12325-022-02345-5. Epub 2022 Oct 29. PMID 36308640